CLINICAL TRIAL: NCT02145676
Title: OnabotulinumtoxinA Treatment in Adult Patients With Upper Limb Spasticity
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-127; 2013-002346-37 (EudraCT Number)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Muscle Spasticity; Stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- onabotulinumtoxinA 500U (Experimental): OnabotulinumtoxinA 500U injected into predefined muscles of the study limb on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- onabotulinumtoxinA 300U (Experimental): OnabotulinumtoxinA 300U injected into predefined muscles of the study limb on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- placebo (normal saline) (Placebo Comparator): Placebo (normal saline) injected into predefined muscles of the study limb on Day 1.
  Interventions: Drug: placebo (normal saline)

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA injected into predefined muscles of the study limb on Day 1.
  Other Names: BOTOX®; botulinum toxin type A
  Arms: onabotulinumtoxinA 300U; onabotulinumtoxinA 500U
Drug: placebo (normal saline) — Placebo (normal saline) injected into predefined muscles of the study limb on Day 1.
  Arms: placebo (normal saline)

SUMMARY:
This is a safety and efficacy study of onabotulinumtoxinA in poststroke patients with upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb spasticity in the elbow and shoulder due to stroke, with the most recent stroke at least 3 months ago

Exclusion Criteria:

* Spasticity in the non-study upper limb that requires treatment
* Presence of fixed contractures in of the study muscles in elbow or shoulder
* Profound atrophy of muscles to be injected
* Previous surgical intervention, nerve block, or muscle block for the treatment of spasticity in the study limb in the last 12 months
* Injection of corticosteroids or anesthetics, use of casting or dynamic splinting or constraint-induced movement therapy (CIMT) for the study limb within 3 months
* Ultrasound therapy, electrical stimulation, or acupuncture in the study limb within 1 month
* Condition other than stroke contributing to upper limb spasticity
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, and/or amyotrophic lateral sclerosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Overland Park, Kansas, United States
- Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Started | 17 | 18 | 18
Completed | 17 | 18 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 17 | 18 | 18 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (11.46) | 59.7 (10.36) | 56.2 (8.30) | 58.2 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 10 | 22
  Male | 13 | 10 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified Ashworth Scale-Bohannon (MAS-B) Score of Elbow Flexors Using a 6-Point Scale
Description: The MAS-B is a 6-point scale used to evaluate spasticity based on grading the resistance encountered in the elbow flexors by passively moving the elbow flexor muscles through their range of motion. The score ranges from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Scores are converted to a 0 to 5 grade. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat: all randomized patients who were analyzed according to randomization assignment, regardless of treatment actually received
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 17 | 18 | 18
Scores on a Scale
  Baseline | 4.12 (0.332) | 4.06 (0.236) | 4.17 (0.383)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 18 | 17
  Change from Baseline at Week 6 | -1.62 (1.455) | -1.47 (1.247) | -0.74 (0.970)

2. Secondary Outcome: Change From Baseline in the MAS-B Score of Shoulder Adductors Using a 6-Point Scale
Description: The MAS-B is a 6-point scale used to evaluate spasticity based on grading the resistance encountered in the shoulder adductors by passively moving the shoulder adductor muscles through their range of motion. The score ranges from 0 (no increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension). Scores are converted to a 0 to 5 grade. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 17 | 18 | 18
Scores on a Scale
  Baseline | 4.00 (0.000) | 4.06 (0.236) | 4.00 (0.000)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 18 | 17
  Change from Baseline at Week 6 | -1.59 (1.263) | -1.39 (1.042) | -1.44 (1.004)

3. Secondary Outcome: Change From Baseline in Pain on an 11-Point Scale
Description: The patient is asked to select a number that best describes his/her pain in the treated areas of the study limb on an 11-point scale from 0 = "no pain" to 10 = "pain as bad as can be imagined". Patients are instructed to recall their average pain in the study limb during the 48-hour period prior to the visit. Patients with a baseline pain score >0 are included in the analyses. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 11 | 10 | 13
Scores on a Scale
  Baseline | 4.89 (2.714) | 6.05 (3.197) | 5.13 (3.586)
  Change from Baseline at Week 6: number analyzed (Participants) | 11 | 10 | 11
  Change from Baseline at Week 6 | -2.08 (3.585) | -2.51 (4.606) | -2.64 (3.857)

4. Secondary Outcome: Change From Baseline in the Dressing Domain Score on the Spasticity Impact Assessment-Upper Limb (SIA-UL)
Description: The SIA-UL asks the patient to assess the impact of upper limb spasticity in his/her daily life on a 19-item scale. The scale covers impacts on activities of dressing, showering/bathing, and self-care. The SIA score ranged from 0 (not at all difficult) to 4 (extremely difficult) for each question. The dressing domain was calculated based on the average of 2 questions.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 17 | 18 | 18
Scores on a Scale
  Baseline | 2.61 (1.346) | 2.91 (1.123) | 2.82 (1.092)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 18 | 17
  Change from Baseline at Week 6 | -0.36 (0.854) | -0.27 (0.932) | -0.55 (1.082)

5. Secondary Outcome: Change From Baseline in the Showering/Bathing Domain Score on the Spasticity Impact Assessment-Upper Limb (SIA-UL)
Description: The SIA-UL asks the patient to assess the impact of upper limb spasticity his/her daily life on a 19-item scale. The scale covers impacts on activities of dressing, showering/bathing, and self-care. The SIA score ranged from 0 (not at all difficult) to 4 (extremely difficult) for each question. The showering/bathing domain was based on a single question.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 17 | 18 | 18
Scores on a Scale
  Baseline | 2.71 (1.231) | 2.69 (1.263) | 2.58 (1.188)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 18 | 17
  Change from Baseline at Week 6 | -0.62 (1.147) | -0.36 (1.247) | -0.51 (1.064)

6. Secondary Outcome: Change From Baseline in the Self-Care Domain Score on the Spasticity Impact Assessment-Upper Limb (SIA-UL)
Description: The SIA-UL asks the patient to assess the impact of upper limb spasticity in his/her daily life on a 19-item scale. The scale covers impacts on activities of dressing, showering/bathing, and self-care. The SIA score ranged from 0 (not at all difficult) to 4 (extremely difficult) for each question. The self-care domain was calculated based on the average of 4 questions.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Number analyzed (Participants) | 17 | 18 | 18
Scores on a Scale
  Baseline | 2.58 (1.234) | 2.61 (1.189) | 2.61 (1.086)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 18 | 17
  Change from Baseline at Week 6 | -0.26 (0.779) | -0.21 (0.667) | -0.48 (1.094)

ADVERSE EVENTS:
Description: The Safety Population included all enrolled patients who received a treatment injection. The Safety Population was used to assess adverse events and serious adverse events.
Arm/Group | onabotulinumtoxinA 500U | onabotulinumtoxinA 300U | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 2/17 | 0/18 | 3/18
Other Adverse Events (participants affected / at risk) | 4/17 | 5/18 | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | onabotulinumtoxinA 500U (N=17) | onabotulinumtoxinA 300U (N=18) | Placebo (Normal Saline) (N=18)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/13 | 0/10 | 0/8
Seizure (Nervous system disorders) | 0 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA 500U (N=17) | onabotulinumtoxinA 300U (N=18) | Placebo (Normal Saline) (N=18)
Bronchitis (Infections and infestations) | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Electromyogram abnormal (Investigations) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.